CLINICAL TRIAL: NCT07163039
Title: The Effect of Dual Task Training on Cognitive in Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Burcu AKKURT, Assistant Professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 63.2025fbu
Record Dates: First submitted 2025-08-21; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Dual-Task Training
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-task motor-cognitive training (Experimental): Participants assigned to this group will undergo dual-task motor-cognitive training, which combines physical exercises with simultaneous cognitive tasks. Sessions will last 45-60 minutes, three times per week, for 8 weeks. Exercises will include gait and balance activities performed while engaging in cognitive tasks such as arithmetic, memory recall, or word association.
  Interventions: Other: Dual-Task Motor-Cognitive Training
- Conventional Exercise Training (Active Comparator): Participants in this group will receive a conventional exercise program focusing on strength, flexibility, and balance without a cognitive component. Sessions will last 45-60 minutes, three times per week, for 8 weeks, and will be supervised by a physiotherapist.
  Interventions: Other: Conventional Exercise Training

INTERVENTIONS:
Other: Dual-Task Motor-Cognitive Training — Participants assigned to this group will undergo dual-task motor-cognitive training, which combines physical exercises with simultaneous cognitive tasks. Sessions will last 45-60 minutes, three times per week, for 8 weeks. Exercises will include gait and balance activities performed while engaging in cognitive tasks such as arithmetic, memory recall, or word association.
  Arms: Dual-task motor-cognitive training
Other: Conventional Exercise Training — Participants in this group will receive a conventional exercise program focusing on strength, flexibility, and balance without a cognitive component. Sessions will last 45-60 minutes, three times per week, for 8 weeks, and will be supervised by a physiotherapist.
  Arms: Conventional Exercise Training

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of dual-task training on cognitive functions in patients with Alzheimer's disease. Participants will be randomly assigned to either a dual-task training group or a conventional exercise group. The intervention will last 8 weeks, with three supervised sessions per week. Cognitive performance, mobility, balance, and quality of life will be assessed before and after the intervention.

DETAILED DESCRIPTION:
Alzheimer's disease is a progressive neurodegenerative disorder characterized by impairments in memory, executive function, and daily activities. Conventional exercise programs may improve mobility and physical performance, but their impact on cognition is limited. Dual-task training, which integrates motor and cognitive activities simultaneously, has emerged as a promising strategy to enhance neuroplasticity and functional independence in individuals with cognitive decline.

In this study, participants diagnosed with Alzheimer's disease according to standard clinical criteria will be recruited. After baseline assessments, participants will be randomly allocated to one of two groups:

Experimental Group (Dual-Task Training): Participants will perform exercises combining cognitive tasks (e.g., arithmetic, memory recall, word association) with simultaneous motor tasks (e.g., walking, balance training, functional mobility exercises).

Control Group (Conventional Exercise): Participants will engage in standard physical exercises focusing on strength, flexibility, and balance, without added cognitive tasks.

The intervention will span 8 weeks, with three 45-60 minute sessions per week, conducted under supervision by a physiotherapist.

Outcome Measures

Primary Outcomes: Cognitive performance assessed by the Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA).

Secondary Outcomes: Functional mobility (Timed Up and Go test), balance (Berg Balance Scale), and quality of life (QoL-AD questionnaire).

Hypothesis

It is hypothesized that dual-task training will lead to greater improvements in cognitive performance and functional independence compared to conventional exercise programs. This study may provide evidence supporting dual-task rehabilitation as a complementary approach in the management of Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Diagnosed with mild-stage Alzheimer's disease (According to DSM-5 or NINCDS-ADRDA criteria)
* MoCA score between 10-25 (Indicating sufficient cognitive capacity for dual-task training)
* Ability to walk independently or with minimal assistance
* Adequate hearing and vision to enable communication
* Physical and mental capacity to participate in the dual-task training protocol
* Provision of written informed consent (signed informed consent form)

Exclusion Criteria:

* Diagnosis of advanced-stage Alzheimer's disease (MoCA < 10)
* Presence of additional neurological disorders affecting the motor system (e.g. Parkinson's disease, stroke, multiple sclerosis)
* Severe hearing or vision impairment (inability to respond to visual or auditory stimuli)
* History of psychiatric disorders (e.g., major depression, schizophrenia)
* Orthopedic or cardiopulmonary conditions that would prevent participation in dual-task training
* Participation in another cognitive or physical rehabilitation program within the last 3 months
* Individuals with unstable cognitive status due to recent medication changes

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
d2 Test of Attention | From enrollment to the end of treatment at 8 weeks
  A widely used neuropsychological test evaluating visual attention and processing speed. Participants are asked to quickly and accurately mark target symbols (e.g., the letter "d" with two dashes) among distractors on a sheet consisting of similar letters and symbols.
Trail Making Test Part A (TMT-A) | From enrollment to the end of treatment at 8 weeks
  Assesses visual attention, processing speed, and psychological flexibility. The participant is required to connect numbered circles from 1 to 25 in order as quickly as possible.
Stroop Test | From enrollment to the end of treatment at 8 weeks
  Stroop Test: Evaluates executive functions and attentional control. The participant must state the ink color of a word rather than reading the written word itself (e.g., the word "Blue" written in red ink should be answered as "red")
Trail Making Test Part B (TMT-B): | From enrollment to the end of treatment at 8 weeks
  Trail Making Test Part B (TMT-B): Used to assess executive functions, cognitive flexibility, and attention. The participant alternates between numbers and letters in sequence (1-A-2-B-3-C…)
Montreal Cognitive Assessment (MoCA) | From enrollment to the end of treatment at 8 weeks
  Montreal Cognitive Assessment (MoCA): Evaluates memory, attention, executive functions, and visuospatial skills. It is a standard and validated tool for monitoring cognitive status and comparing pre- and post-intervention performance in Alzheimer's patients

SECONDARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) | From enrollment to the end of treatment at 8 weeks
  Symbol Digit Modalities Test (SDMT): Measures processing speed and attention. Participants are presented with a key of symbol-digit pairings and asked to match as many symbols with their corresponding digits as possible within a set time
Functional Near-Infrared Spectroscopy (fNIRS) | From enrollment to the end of treatment at 8 weeks
  Functional Near-Infrared Spectroscopy (fNIRS): A non-invasive method to measure prefrontal cortex activation by monitoring oxygenated and deoxygenated hemoglobin levels
Disability Assessment for Dementia (DAD) | From enrollment to the end of treatment at 8 weeks
  Disability Assessment for Dementia (DAD): Developed to assess independence in activities of daily living among individuals with dementia. It evaluates both basic and instrumental activities of daily living, including self-care and social functioning
Dual Task Protocol | From enrollment to the end of treatment at 8 weeks
  Dual Task Protocol: Participants will perform physical and cognitive tasks simultaneously. For example, during walking, they will be asked to complete word generation, simple arithmetic, or other attention-demanding tasks
Performance Measures: Walking speed | From enrollment to the end of treatment at 8 weeks
  Walking speed (measured using a metronome or gait analysis system).
Performance Measures: Step count | From enrollment to the end of treatment at 8 weeks
  Step count (measured using a metronome or gait analysis system).
Performance Measures: Number of correct response Number of correct responses | From enrollment to the end of treatment at 8 weeks
  Number of correct responses recorded during the secondary cognitive task.
Performance Measures: incorrect response | From enrollment to the end of treatment at 8 weeks
  Percentage of incorrect responses recorded during the secondary cognitive task.
Gait Analysis System: Walking speed during single-task walking | From enrollment to the end of treatment at 8 weeks
  Provides objective evaluation of walking dynamics using pressure sensors, motion capture systems, or accelerometers.
Gait Analysis System: Step length during single-task walking | From enrollment to the end of treatment at 8 weeks
  Provides objective evaluation of walking dynamics using pressure sensors, motion capture systems, or accelerometers.
Gait Analysis System:Balance during dual-task walking | From enrollment to the end of treatment at 8 weeks
  Provides objective evaluation of walking dynamics using pressure sensors, motion capture systems, or accelerometers.
Gait Analysis System: Postural control during dual-task walking | From enrollment to the end of treatment at 8 weeks
  Provides objective evaluation of walking dynamics using pressure sensors, motion capture systems, or accelerometers.
Electromyography (EMG) | From enrollment to the end of treatment at 8 weeks
  Electromyography (EMG): Measures muscle electrical activity through surface electrodes, providing data on contraction duration, activation levels, and coordination (De Luca, 1997). EMG will be used to assess changes in motor control and muscle activation during dual-task training.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye AKÇAY, PhD, Principal Investigator — Fenerbahçe University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT07163039/Prot_SAP_000.pdf